CLINICAL TRIAL: NCT01902186
Title: Switching HIV-positive Women on Tenofovir/Emtricitabine Plus Boosted Atazanavir to RALtegravir Plus Boosted ATazanavir: A Pilot Randomized Clinical Trial Investigating 48-weeks Changes in Bone Mineral Density
Brief Title: Bone Mineral Density Changes in HIV-positive Females With Osteopenia Switching to Raltegravir
Acronym: RALBAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Giovanni Di Perri (Other)
Collaborators: University of Turin, Italy (Other); University of Milan (Other)
Responsible Party: Sponsor-Investigator, Giovanni Di Perri, Full professor of Infectious Diseases, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RALBAT
Record Dates: First submitted 2013-07-10; First posted 2013-07-18 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: HIV Infection; Osteopenia
Keywords: HIV; osteopenia; t-score; DEXA; tenofovir; raltegravir
MeSH Terms: conditions — HIV Infections; Bone Diseases, Metabolic | interventions — Raltegravir Potassium; Atazanavir Sulfate; Ritonavir; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- raltegravir (Experimental): raltegravir and atazanavir and ritonavir
  Interventions: Drug: raltegravir and atazanavir and ritonavir
- tenofovir/emtricitabine (Active Comparator): tenofovir/emtricitabine and atazanavir and ritonavir
  Interventions: Drug: tenofovir/emtricitabine and atazanavir and ritonavir

INTERVENTIONS:
Drug: raltegravir and atazanavir and ritonavir — switch tenofovir/emtricitabine to raltegravir
  Other Names: Isentress (raltegravir); Reyataz (atazanavir); Norvir (ritonavir)
  Arms: raltegravir
Drug: tenofovir/emtricitabine and atazanavir and ritonavir — no change in antiretroviral treatment; patients will continue their regimen (tenofovir/emtricitabine and atazanavir and ritonavir)
  Other Names: tenofovir/emtricitabine (Truvada); atazanavir (Reyataz); ritonavir (norvir)
  Arms: tenofovir/emtricitabine

SUMMARY:
Given the high prevalence of bone alteration in the course of HIV infection or antiretroviral treatment and the favourable properties of raltegravir the investigators designed this pilot randomized and controlled study. Adult female HIV-positive patients on successful treatment with tenofovir/emtricitabine plus atazanavir plus ritonavir will be randomized either to continue such a regimen or to switch to raltegravir plus atazanavir plus ritonavir. Bone mineral density changes will be compared in the two groups at 48 weeks: the hypothesis is that removing tenofovir and using tenofovir will increase bone mineral density at 48 weeks.

DETAILED DESCRIPTION:
The objective is to assess the improvement in Bone Mineral Density and markers of bone turnover in women on TDF/FTC (tenofovir disoproxil fumarate/ emtricitabine)+ ATV/r (atazanavir/ritonavir) in a switch arm (RAL (raltegravir) + ATV/r) vs. an unchanged arm (TDF/FTC + ATV/r).

The clinical hypothesis is that removing tenofovir (associated to a boosted PI, and therefore in the worst clinical scenario) in both pre-menopausal and menopausal women could be beneficial and being associated with reduced bone mineral density loss measured by DEXA (densitometry)scan scores and markers of bone turnover. The underlying mechanism is believed to be the reduction in hyper-phosphaturia induced by proximal tubular dysfunction: therefore measuring renal tubular markers and hormones involved in calcium and phosphorus homeostasis (such as vitamin D and parathormone) will explain the suspected mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Adult HIV-positive female patients;
* osteopenia (t-score from -1 to -2.5);
* On antiretroviral treatment with tenofovir/emtricitabine and atazanavir/ritonavir (300/100 mg) for at least six months;
* Plasma HIV RNA below 50 copies/ml since six months;
* Premenopausal women: female patients at any phase of the reproductive period with regular menstrual cycles and normal FSH (< 25 ng/mL) That would probably exclude patients with ovarian or endocrinological dysfunctions. Pre and postmenopausal should be therefore well-characterized.
* Women in menopausal period (the menopause was defined as 12 months of amenorrhoea without any pathological or physiological cause and using the endocrinological definition of ovary insufficiency (LH (Luteic hormone) >25ng/mL, FSH (follicule stimulating hormone)>25ng/mL and E2 (Estradiol)<30ng/mL).
* Each premenopausal sexually active subject of child-bearing potential must agree to use a medically accepted method of contraception while receiving protocol-specified medication and for 3 months after stopping the medication.Medically accepted methods of contraception include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD (intrauterine device), inert or copper-containing IUD, hormone-releasing IUD, systemic hormonal contraceptive, and surgical sterilization (eg, hysterectomy or tubal ligation).
* Postmenopausal women are not required to use contraception.

Exclusion Criteria:

* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate.
* Documented resistance to Raltegravir or/and Atazanavir.
* Patient with significant hypersensitivity or other contraindication to any of the components of the study drugs.
* Patient has a current (active) diagnosis of acute hepatitis due to any cause
* Patient with coinfection HIV/HBV (Human Hepatitis virus B)
* Liver cirrhosis
* Osteoporosis (t-score less than 2.5).
* Secondary endocrinological cause of low BMD (Bone mineral density)
* Chronic steroid intake;
* Chronic kidney disease (estimated glomerular filtration rate below 60 ml/min);
* Concomitant use of bisphosphonate.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Variations from baseline in DEXA-measured bone mineral density (t-score, spine and femur) | 48 weeks

SECONDARY OUTCOMES:
variations from baseline in CTX (C-terminal telopeptide of type I collagen) and OC (Osteocalcin) | 24 and 48 weeks
To assess the variation in renal function | 48 weeks
  glomerular filtration rate, urinary markers of tubular dysfunction (nondiabetic glucosuria, altered resorption of phosphorus, hyperaminoaciduria, b2-micro-globuline excretion and abnormal uric acid excretion.) and urinary retinol binding protein

OTHER OUTCOMES:
Cholesterol changes at 48 weeks in the two arms | 48 weeks
  Changes in Cholesterol levels in the two arms
Triglycerides changes in the two arms | 48 weeks
  Changes in Tryglicerdies levels in the two arms
Glucose Fasting Levels changes in the two arms | 48 weeks
  Changes in Glucose Fasting Levels in the two arms
Insulin changes in the two arms | 48 weeks
  Changes in Insulin levels in the two arms
Parathyroid hormone changes in the two arms | 48 weeks
  Changes in Parathyroid hormone levels in the two arms
Vitamine D (25-OH-Vitamine D) changes in the two arms | 48 weeks
  Changes in Vitamine D (25-OH-Vitamine D)levels in the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Di Perri, MD, PhD, Principal Investigator — University of Turin, Italy
Locations (2):
- Italy (2):
  - University of Milano, Milan
  - University of Torino, Torino